CLINICAL TRIAL: NCT04892433
Title: Tissue Study in Patients Undergoing CAR-T Cell Therapy
Brief Title: Tissue Study in Patients Undergoing CAR-T Cell Therapy (CAR_21_01)
Acronym: CAR_21_01
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, Hematologist Doctor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CAR_21_01
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: CAR-T Therapy Complications
Keywords: DNA-methylation; CAR-T Therapy; microRNA; lymphocyte and myeloid populations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The "CAR-T" immunotherapy ("Chimeric Antigen Receptor T cell therapies") is a therapy based on T cells expressing a chemical receptor for a specific antigen indicated for patients with some types of oncohematological pathologies that have not responded to other forms treatment, such as: relapsed or refractory non-Hodgkin's lymphomas, including diffuse large B-cell lymphoma, primary B-cell mediastinal lymphoma, transformed follicular lymphoma, mantle cell lymphoma, acute lymphoblastic leukemia, in children and young adults (<26 years) and multiple myeloma. This therapy is an absolutely innovative approach which consists of a personalized live cell immunotherapy that modifies the immune system of the recipient patient to make it able to recognize and eradicate the neoplastic cells expressing the antigen towards which the cells have been engineered.

This approach has several biological advantages:

1. to supply the patient with "reprogrammed T cells" with a new and specific activation mechanism;
2. overcoming immune tolerance towards cancer cells;
3. bypassing HLA-mediated antigen recognition restriction mechanisms;

DETAILED DESCRIPTION:
The "CAR-T" immunotherapy ("Chimeric Antigen Receptor T cell therapies") is a therapy based on T cells expressing a chemical receptor for a specific antigen indicated for patients with some types of oncohematological pathologies that have not responded to other forms treatment, such as: relapsed or refractory non-Hodgkin's lymphomas, including diffuse large B-cell lymphoma, primary B-cell mediastinal lymphoma, transformed follicular lymphoma, mantle cell lymphoma, acute lymphoblastic leukemia, in children and young adults (<26 years) and multiple myeloma. This therapy is an absolutely innovative approach which consists of a personalized live cell immunotherapy that modifies the recipient patient's immune system to make it able to recognize and eradicate the neoplastic cells expressing the antigen towards which the cells have been engineered. CAR-T therapy uses specific immune cells (T lymphocytes) of the patient, isolated from his peripheral blood, engineered through the integration of genetic material encoding the chimeric receptor, expanded in vitro and then re-infused to activate the immune system response against the disease.

This approach has several biological advantages:

1. to supply the patient with "reprogrammed T cells" with a new and specific activation mechanism;
2. overcoming immune tolerance towards cancer cells;
3. bypassing HLA-mediated antigen recognition restriction mechanisms; The CAR-T therapies that have obtained the Marketing Authorization (AIC) in the European Union and in Italy are: the drug Kymriah, drug Yescarta.

The therapeutic indications for which they have been approved are:

* Kymriah (tisagenlecleucel): pediatric and young adult patients up to 25 years of age with B-cell acute lymphoblastic leukemia who have never responded to chemotherapy, or who have relapsed after allogeneic haematopoietic stem cell transplantation or after at least 2 lines chemotherapy; patients with diffuse large B cell lymphoma or DLBCL who have already undergone at least 2 lines of systemic therapy;
* Yescarta (axicabtagene ciloleucel): patients with diffuse large B cell lymphoma or DLBCL, primary mediastinal B cell lymphoma or PMBCL who have already received at least 2 lines of systemic therapy. CAR-T therapies represent an important therapeutic option for the lymphoproliferative diseases listed above and have been studied in patients in whom previous standard strategies (chemotherapy and haematopoietic stem cell transplantation) have not proved effective.

Although they represent an effective last therapeutic option in patients with advanced disease and resistant to traditional chemotherapy lines, the use of CAR-T therapies is not without serious complications, quite the contrary. In particular, there are:

* Cytokine Release Syndrome (CRS);
* Reduction of B lymphocytes (hypogammaglobulinemia);
* Neurological adverse reactions;

Understanding of the determinants of the massive inflammatory response underlying the toxicity of CAR-T therapy remains largely unclear. It is a shared opinion in the medical-scientific community that what is defined as the "target effect" of CAR cells on target tumor cells, and the consequent immune response, is one of the factors triggering a massive pro-inflammatory cytokine reaction, but the mechanisms that are the basis and that they can predict and personalize the treatment, or even prevent it, are not yet defined. It is hypothesized, and several studies are beginning to be available in this regard, that the composition and ratios of leukocyte populations (CD4 and CD8 among others) used for the production of CAR T may influence the clinical outcome in the patient. In particular, the proliferation and persistence of CAR cells in the patient are key factors in determining the effectiveness of the therapy itself. Hence the need to characterize the various cell subsets both in the CD3 + CAR + population and in the CD3 + CAR- population in the patient's clinical course. It is also fundamental to study the epigenetic status of the lymphocyte populations themselves, as well as the biological age of the patient connected to it. It is in fact an element that is believed to play a fundamental role in the clinical response. In fact, the assessment of the biological age of a subject is an index composed of molecular markers (such as the epigenetic status of nucleated cells), strongly correlated with the chronological age, but capable of expressing the speed of aging of the single individual, as well as of the cells of his immune system, and consequently capable of highlighting with greater emphasis than the chronological age the health risks associated with the therapy and his inflammatory state. A further element to consider in the overall picture we are considering is the role that microRNAs (miRNAs) play as crucial regulators of T-cell survival, differentiation and function, all of which are key factors influencing the outcome of immunotherapy. adoptive based on CAR cells. MicroRNAs are short strands of RNA with a regulatory function of cellular gene expression, especially in the modulation of inflammation. For this reason, the study of them in the context we are considering is of primary importance.

Given these premises, the primary objectives of the study are the following:

1. Study of epigenetics in peripheral blood samples taken from patients undergoing CAR-T therapy. In particular, the epigenetic analysis will be carried out in the circulating leukocyte and extracellular fraction contained in the plasma nanovesicles in order to determine the epigenome and its correlation with the clinical outcome of the patients;
2. Study of microRNAs extracted from extracellular vesicles and leukocytes of patients undergoing CAR-T therapy in order to correlate the levels with the clinical outcome of patients;
3. Study of lymphocyte and myeloid populations in the haematological patient PRE and POST CAR-T cell infusion in order to correlate the levels with the clinical outcome of the patients; To pursue these objectives, a monocentric and exploratory study will be launched, which involves the use of human tissues in vitro, in this case blood, in patients subjected to infusion of CAR-T cells. The study will be offered to all patients undergoing CAR-T cell infusion at the Advanced Cell Therapy Program of the IRCCS University Hospital of Bologna. The study is expected to last 5 years with an enrollment of 35 patients per year. The analysis of the samples will be carried out in the laboratories of Prof Massimiliano Bonafè, co-author of the study, free of charge.

Peripheral blood samples will be used to carry out the study and will be taken at the following times:

* to apheresis;
* upon entering the ward;
* on day -1;
* on day 0 (2 hours post-infusion);
* per day +1, +3, +5, +7, +9, +11, +13, +30, +90, +180, +365;

The sampling of tissues coincides with the sampling that represent the current standard in routine clinical practice in the transplanted patient; therefore the samples will be obtained taking care not to invalidate the normal diagnostic-assistance procedures. The results of this study will have a clinical-care impact of primary importance aimed at managing the complications of CAR-T therapy and at understanding the biological mechanisms underlying them.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 years. Patients with haematological pathology admitted to be subjected to CAR-T Therapy at the Advanced Cell Therapy Program, IRCCS University Hospital of Bologna.

Patients who consent to participate in this study after signing informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nell'ambito del normale percorso assistenziale verranno arruolati tutti i pazienti ammessi a essere sottoposti a CAR-T Therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Study of epigenetics | 5 years
  Study of epigenetics in peripheral blood samples taken from patients undergoing CAR-T therapy. In particular, the epigenetic analysis will be performed in the circulating leukocyte and extracellular fraction contained in the plasma nanovesicles in order to determine the epigenome and its correlation with the clinical outcome.
Study of microRNA | 5 years
  study of microRNAs extracted from extracellular vesicles and leukocytes of patients undergoing CAR-T therapy in order to correlate levels with clinical outcome.
study of lymphocyte and myeloid populations | 5 years
  study of lymphocyte and myeloid populations in the haematological patient PRE and POST CAR-T cell infusion in order to correlate the levels with the clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bonifazi, MD, Principal Investigator — Advanced Cell Therapy Program, IRCCS University Hospital of Bologna
Locations (1):
- IRCC, University Hospital of Bologna, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Matteis S, Dicataldo M, Casadei B, Storci G, Laprovitera N, Arpinati M, Maffini E, Cortelli P, Guarino M, Vaglio F, Naddeo M, Sinigaglia B, Zazzeroni L, Guadagnuolo S, Tomassini E, Bertuccio SN, Messelodi D, Ferracin M, Bonafe M, Zinzani PL, Bonifazi F. Peripheral blood cellular profile at pre-lymphodepletion is associated with CD19-targeted CAR-T cell-associated neurotoxicity. Front Immunol. 2023 Jan 16;13:1058126. doi: 10.3389/fimmu.2022.1058126. eCollection 2022. PMID 36726971